CLINICAL TRIAL: NCT01373112
Title: Articulating Versus Static Antibiotic Loaded Spacers for the Treatment of Prosthetic Knee Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: Central DuPage Hospital (Other); Joint Implant Surgeons, Inc. (Other); Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Peter N. Chalmers, MD, Resident, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPACERKNEE
Record Dates: First submitted 2011-06-06; First posted 2011-06-14 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Osteoarthritis; Knee Infection; Prosthetic Joint Infection; Complications; Arthroplasty, Infection or Inflammation; Complications; Arthroplasty
Keywords: arthroplasty; knee replacement; Osteoarthritis; knee Infection; Prosthetic Joint Infection; Complications; Arthroplasty, Infection or Inflammation; Complications; Arthroplasty
MeSH Terms: conditions — Osteoarthritis; Infections; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Static Spacer (Experimental): After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or a static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of the infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed of 3 g of Vancomycin and 1 g of Tobramycin for each 40 g packet of cement. Static spacers will be hand-made to fit the femoral and tibial exposed metaphyses as a solid block with associated antibiotic cement coated tibial and femoral intramedullary rod, such that knee motion will be minimized.
  Interventions: Procedure: Static Spacer
- Articulating Spacer (Experimental): After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or a static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of the infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed of 3 g of Vancomycin and 1 g of Tobramycin for each 40 g packet of cement. Articulating spacers will be formed of antibiotic impregnated cement using the Stage One system (Biomet, Warsaw, IN).
  Interventions: Procedure: Articulating Spacer

INTERVENTIONS:
Procedure: Static Spacer — After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or a static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of the infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed of 3 g of Vancomycin and 1 g of Tobramycin for each 40 g packet of cement. Static spacers will be hand-made to fit the femoral and tibial exposed metaphyses as a solid block with associated antibiotic cement coated tibial and femoral intramedullary rod, such that knee motion will be minimized.
  Arms: Static Spacer
Procedure: Articulating Spacer — After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or a static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of the infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed of 3 g of Vancomycin and 1 g of Tobramycin for each 40 g packet of cement. Articulating spacers will be formed of antibiotic impregnated cement using the Stage One system (Biomet, Warsaw, IN).
  Arms: Articulating Spacer

SUMMARY:
Infection remains a difficult-to-treat complication of total knee arthroplasty. The gold standard treatment is two-stage removal of the prosthesis with later replacement of permanent implants. The first stage consists of removal of the infected arthroplasty components and the surrounding devitalized tissue, copious pulsed irrigation, and placement of a temporary antibiotic-impregnated cement spacer. This spacer typically is left in place six weeks, during which time the patient receives intravenous antibiotics. After the surgeon feels that the infection has been eradicated, or if the patient requires repeat debridement, a second operative procedure is performed. While the use of an antibiotic-loaded spacer is well accepted, whether the spacer should immobilize the knee (a so-called "static" spacer) or allow for range of motion (a so-called "articulating" spacer) is controversial. Proponents of articulating spacers argue that they prevent scarring of the musculature surrounding the knee resulting in easier reimplantation, improved long-term knee function, and improved range of motion. Proponents of static spacers argue that immobilization of the periarticular soft tissues aids in clearance of the infection and is simpler to fashion intraoperatively. While good results have been described with both methods, comparative trials have been conflicting as to whether spacer design alters knee function, operative time, and range of motion. Equipoise exists within the literature, and no randomized clinical trial has been conducted to evaluate this issue.

The purpose of this study is to compare articulating and static antibiotic-impregnated spacers for the treatment of chronic periprosthetic infection complicating total knee arthroplasty through a prospective, randomized clinical trial. The goals of this trial are to determine the effect of spacer design upon eradication of infection, knee function, ease of reimplantation, and range of motion. The investigators hypothesize that articulating spacers will provide shorter operative times at reimplantation, while improving knee function and range of motion.

DETAILED DESCRIPTION:
After diagnosis of infection and informed consent, patients will be taken to the operating room. After anesthetization, patients will be randomized to either an articulating spacer or a static spacer. Randomization will be performed by prepared opaque envelopes administered by a nonparticipant in the study. After a complete debridement of devitalized tissue, explantation of the infected components and any associated cement, either an articulating or static spacer will be placed. All spacers will be formed of 3 g of Vancomycin and 1 g of Tobramycin for each 40 g packet of cement. Articulating spacers will be formed of antibiotic impregnated cement using the Stage One system (Biomet, Warsaw, IN). Static spacers will be hand-made to fit the femoral and tibial exposed metaphyses as a solid block with associated antibiotic cement coated tibial and femoral intramedullary rod, such that knee motion will be minimized.

Post-operatively, all patients will be made touch-down weight bearing protected with a walker or crutches. If a static spacer is placed, patients will be immobilized using with a knee immobilizer. If an articulating spacer is utilized, range of motion will be allowed to the limits of stability as determined in the operating room and protected with a hinged knee brace. At the time of reoperation, the joint will be aspirated and multiple cultures obtained along with intraoperative histopathological analysis to evaluate for persistent infection.

Data collected preoperatively will include age, gender, laterality, etiology of knee degeneration, comorbidities, Knee Society score, and infecting organisms. The Knee Society score has been used extensively in the study of revision knee arthroplasty and has been found to be reliable and valid and will be determined pre-operatively and at all follow-up visits.

Data collected at the time of implant removal and reimplantation will include operative time, blood loss, and need for an extensile exposure. Radiographs performed immediately following and just prior to reimplantation will be reviewed to determine if the spacer utilized has caused bone loss; bone loss to the cut bony surfaces will be confirmed intraoperatively. At each follow-up visit radiographic appearance, the Knee Society Score, knee range of motion, recurrence of infection, and the need for revision or reoperation of any kind on the knee will be determined.

All portions of this study will be part of conventional care except for randomization to either a static or articulating spacer. Which type of spacer is used currently depends upon the judgment of the attending surgeons and both are used routinely.

The primary outcome variable will be range of motion. A power analysis was conducted with the assistance of Dr. Mario Moric at Rush using range of motion as our primary outcome variable, with standard deviations culled from two of the largest series to date -Van Thiel and colleagues (2010) and Fehring and colleagues (2000). For an 80% chance of detecting a predetermined clinically significant difference of 10 degrees, 53 patients per group, 106 patients total, will be needed. To account for attrition, our target sample size will be 140 patients.

ELIGIBILITY:
Inclusion Criteria:

1) Diagnosis of a periprosthetic joint infection of a primary total knee arthroplasty with a planned two-stage exchange procedure.

Exclusion Criteria:

1. Infection of a revision as opposed to a primary total knee arthroplasty
2. Medically unfit for operative intervention
3. Extensive bone loss preventing the use of an articulating spacer
4. Soft tissue defects that prevent the use of an articulating spacer
5. Known allergy to polymethylmethacrylate, tobramycin or vancomycin.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2011-12; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Range of motion | Outcomes will be collected until 2 years post-operatively.

SECONDARY OUTCOMES:
Knee Society Score | Outcomes will be collected until 2 years post-operatively.
Operative time | Outcomes will be collected until 2 years post-operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chalmers, MD, Principal Investigator — Rush University Medical Center; Craig Della Valle, MD, Principal Investigator — Rush University Medical Center; Scott Sporer, MD, Principal Investigator — Rush University Medical Center; Adolph Lombardi, MD, Principal Investigator — Joint Implant Surgeons, Inc.; Keith Berend, MD, Principal Investigator — Joint Implant Surgeons, Inc.; Matt Austin, MD, Principal Investigator — Thomas Jefferson Hospital
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Gooding CR, Masri BA, Duncan CP, Greidanus NV, Garbuz DS. Durable infection control and function with the PROSTALAC spacer in two-stage revision for infected knee arthroplasty. Clin Orthop Relat Res. 2011 Apr;469(4):985-93. doi: 10.1007/s11999-010-1579-y. PMID 20878287
- [Background] Haleem AA, Berry DJ, Hanssen AD. Mid-term to long-term followup of two-stage reimplantation for infected total knee arthroplasty. Clin Orthop Relat Res. 2004 Nov;(428):35-9. doi: 10.1097/01.blo.0000147713.64235.73. PMID 15534516
- [Background] Van Thiel GS, Berend KR, Klein GR, Gordon AC, Lombardi AV, Della Valle CJ. Intraoperative molds to create an articulating spacer for the infected knee arthroplasty. Clin Orthop Relat Res. 2011 Apr;469(4):994-1001. doi: 10.1007/s11999-010-1644-6. PMID 21042896
- [Background] Cuckler JM. The infected total knee: management options. J Arthroplasty. 2005 Jun;20(4 Suppl 2):33-6. doi: 10.1016/j.arth.2005.03.004. PMID 15991126
- [Background] Goldman RT, Scuderi GR, Insall JN. 2-stage reimplantation for infected total knee replacement. Clin Orthop Relat Res. 1996 Oct;(331):118-24. doi: 10.1097/00003086-199610000-00016. PMID 8895627
- [Background] Hirakawa K, Stulberg BN, Wilde AH, Bauer TW, Secic M. Results of 2-stage reimplantation for infected total knee arthroplasty. J Arthroplasty. 1998 Jan;13(1):22-8. doi: 10.1016/s0883-5403(98)90071-7. PMID 9493534
- [Background] Emerson RH Jr, Muncie M, Tarbox TR, Higgins LL. Comparison of a static with a mobile spacer in total knee infection. Clin Orthop Relat Res. 2002 Nov;(404):132-8. doi: 10.1097/00003086-200211000-00023. PMID 12439251
- [Background] Fehring TK, Odum S, Calton TF, Mason JB. Articulating versus static spacers in revision total knee arthroplasty for sepsis. The Ranawat Award. Clin Orthop Relat Res. 2000 Nov;(380):9-16. doi: 10.1097/00003086-200011000-00003. PMID 11064968
- [Background] Freeman MG, Fehring TK, Odum SM, Fehring K, Griffin WL, Mason JB. Functional advantage of articulating versus static spacers in 2-stage revision for total knee arthroplasty infection. J Arthroplasty. 2007 Dec;22(8):1116-21. doi: 10.1016/j.arth.2007.04.009. PMID 18078879
- [Background] Hsu YC, Cheng HC, Ng TP, Chiu KY. Antibiotic-loaded cement articulating spacer for 2-stage reimplantation in infected total knee arthroplasty: a simple and economic method. J Arthroplasty. 2007 Oct;22(7):1060-6. doi: 10.1016/j.arth.2007.04.028. PMID 17920482
- [Background] Jamsen E, Sheng P, Halonen P, Lehto MU, Moilanen T, Pajamaki J, Puolakka T, Konttinen YT. Spacer prostheses in two-stage revision of infected knee arthroplasty. Int Orthop. 2006 Aug;30(4):257-61. doi: 10.1007/s00264-006-0102-2. Epub 2006 Mar 25. PMID 16565839
- [Background] Haddad FS, Masri BA, Campbell D, McGraw RW, Beauchamp CP, Duncan CP. The PROSTALAC functional spacer in two-stage revision for infected knee replacements. Prosthesis of antibiotic-loaded acrylic cement. J Bone Joint Surg Br. 2000 Aug;82(6):807-12. doi: 10.1302/0301-620x.82b6.10486. PMID 10990301
- [Background] Hart WJ, Jones RS. Two-stage revision of infected total knee replacements using articulating cement spacers and short-term antibiotic therapy. J Bone Joint Surg Br. 2006 Aug;88(8):1011-5. doi: 10.1302/0301-620X.88B8.17445. PMID 16877598
- [Background] Hofmann AA, Kane KR, Tkach TK, Plaster RL, Camargo MP. Treatment of infected total knee arthroplasty using an articulating spacer. Clin Orthop Relat Res. 1995 Dec;(321):45-54. PMID 7497685
- [Background] Meek RM, Dunlop D, Garbuz DS, McGraw R, Greidanus NV, Masri BA. Patient satisfaction and functional status after aseptic versus septic revision total knee arthroplasty using the PROSTALAC articulating spacer. J Arthroplasty. 2004 Oct;19(7):874-9. doi: 10.1016/j.arth.2004.06.028. PMID 15483804
- [Background] Calton TF, Fehring TK, Griffin WL. Bone loss associated with the use of spacer blocks in infected total knee arthroplasty. Clin Orthop Relat Res. 1997 Dec;(345):148-54. PMID 9418632
- [Background] Fehring TK, Calton TF, Griffin WL. Cementless fixation in 2-stage reimplantation for periprosthetic sepsis. J Arthroplasty. 1999 Feb;14(2):175-81. doi: 10.1016/s0883-5403(99)90122-5. PMID 10065723
- [Background] Asif S, Choon DS. Midterm results of cemented Press Fit Condylar Sigma total knee arthroplasty system. J Orthop Surg (Hong Kong). 2005 Dec;13(3):280-4. doi: 10.1177/230949900501300311. PMID 16365492
- [Background] Ghanem E, Pawasarat I, Lindsay A, May L, Azzam K, Joshi A, Parvizi J. Limitations of the Knee Society Score in evaluating outcomes following revision total knee arthroplasty. J Bone Joint Surg Am. 2010 Oct 20;92(14):2445-51. doi: 10.2106/JBJS.I.00252. PMID 20962195
- [Background] Insall JN, Dorr LD, Scott RD, Scott WN. Rationale of the Knee Society clinical rating system. Clin Orthop Relat Res. 1989 Nov;(248):13-4. PMID 2805470
- [Background] Liow RY, Walker K, Wajid MA, Bedi G, Lennox CM. The reliability of the American Knee Society Score. Acta Orthop Scand. 2000 Dec;71(6):603-8. doi: 10.1080/000164700317362244. PMID 11145388